CLINICAL TRIAL: NCT02313545
Title: Phase I-B Study to Evaluate the Safety, Tolerability and Efficacy of IZN-6NVS for the Treatment of Atrophic Vaginitis or Desquamative Inflammatory Vaginitis
Brief Title: Phase I-B Study to Evaluate the Safety, Tolerability and Efficacy of IZN-6NVS for the Treatment of AV and DIV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Izun Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAV-MAE-101-IL
Record Dates: First submitted 2014-12-07; First posted 2014-12-10 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Atrophic Vaginitis
MeSH Terms: conditions — Atrophic Vaginitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental - IZN-6NVS Cream (Experimental): Eligible women of 3 groups will be assigned to receive IZN-6NVS (IP) - 2.5 g of cream/day for the first 14 days, followed by 3 applications per week for the next 4 weeks.
  Interventions: Drug: IZN-6NVS Cream

INTERVENTIONS:
Drug: IZN-6NVS Cream — IZN-6NVS, a hydrocream containing three herbal extracts, is a polymolecular agent derived from botanical sources. It is composed of a blend of three herbal extracts, Centella asiatica, Echinacea purpurea, and Sambucus nigra.
  Cream concentration: 5%

SUMMARY:
In this open label study, 50 eligible women will be assigned to receive the investigational product (IZN-6NVS) - 2.5 g of cream/day for 14 days, followed by 3 applications per week for the next 4 weeks. Clinical assessment of the severity of vaginitis will be performed at baseline and after 2 and 6 weeks of treatment.

The study will evaluate safety, tolerability and efficacy of IZN-6NVS vaginal cream, in the treatment of atrophic vaginitis (AV) and desquamative inflammatory vaginitis (DIV).

DETAILED DESCRIPTION:
This will be a Phase IB study comprised of three study groups:

* Group 1: Women who are naturally or surgically menopausal and symptomatic for AV, but who decline treatment with topical or systemic estrogen.
* Group 2: Women rendered menopausal as a result of pharmacologic treatment (including, but not limited to, aromatase inhibitor treatment, selective estrogen receptor modifiers (SERMs), and GnRH analog treatment), who decline treatment with topical or systemic estrogen.
* Group 3: Pre-menopausal women diagnosed with DIV.

The study will evaluate safety, tolerability and efficacy of IZN-6NVS vaginal cream, in the treatment of atrophic vaginitis (AV) and desquamative inflammatory vaginitis (DIV).

20 eligible women of groups 1 and 2 and up to 10 eligible women of group 3 will be assigned to receive 2.5 g of cream/day for the first 14 days, followed by 3 applications per week for the next 4 weeks. Clinical assessment of the severity of vaginitis will be performed at baseline and after 2 and 6 weeks of treatment, which will be the end of the study. Patient reported symptom severity will be assessed by questionnaire at baseline and after 2 and 6 weeks of treatment, and at follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Women over age 18
2. For groups 1 and 2:

   I. Self-reported amenorrhea for at least 12 months or documentation of menopause based on serum E2 ≤ 150 pg/ml.

   II. Self-reporting of at least one moderate to severe symptom of vaginal atrophy on a 4-point scale (0=none; 1=mild; 2=moderate; 3=severe):
   * Vaginal dryness
   * Vaginal discomfort or irritation
   * Vaginal itching
   * Vaginal pain associated with sexual activity
   * Vaginal discharge
   * Vaginal Malodor III. Clinical impression of atrophy based on examination of vaginal cytological smear.

   IV. Vaginal pH >4.5

   V. Endometrial thickness ≤5 mm as determined by US, with no abnormalities noted.
3. For group 3 (DIV): Clinical diagnosis of DIV in pre-menopausal women without estrogen deficiency.
4. For all groups:

I. Willing to comply with use of an intravaginal cream containing S. nigra, C. asiatica, and E. purpurea extracts.

II. Normal PAP smear within the last 3 years. III. Able to provide informed consent. -

Exclusion Criteria:

1. Subjects recruited in group 1 should not be actively treated for breast, uterine or ovarian cancer within the past year.
2. Vaginal bleeding of unknown cause within 60 days of enrollment
3. Vaginal infection requiring treatment within 30 days of enrollment
4. Any known allergy to the plant extracts in the study cream
5. Any serious disease; concomitant steroid use or sex hormone treatment
6. Endometrial thickness > 5 mm measured by ultrasound for women enrolled with diagnosis of atrophic vaginitis
7. Use of any vaginal moisturizer (e.g. Replens, Gynomonal) within 30 days of enrollment.
8. In groups 1 and 2, Use of any oral, transdermal, vaginal, or systemic estrogen or estrogen/progestin product within 30 days of enrollment.
9. Current urinary tract infection (UTI) (clinical complaints of UTI or dipstick urinalysis positive for nitrates or blood)
10. History of venous thromboembolic disease.
11. Use of another investigational agent within 12 weeks of screening.
12. Any medical or psychiatric condition that, in the investigator's opinion, would preclude the subject from complying with the study protocol, including the completion of questionnaires.
13. Subjects with DIV who are pregnant or trying to become pregnant will not be included in the study. Similarly, if a subject with DIV becomes pregnant during the study, that patient will be removed from the study.

    -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Safety basis of the following parameters: - General Toxicity: Vital signs (temperature, blood pressure, pulse rate, respiratory rate). - Adverse events and toxicity | 6 weeks
  Safety and tolerability will be evaluated on the basis of the following parameters:
  * General Toxicity: Vital signs (temperature, blood pressure, pulse rate, respiratory rate).
  * Adverse events and toxicity
Change in composite score of vaginal symptoms as assessed by subject questionnaire from baseline | Day 0, Day 14, Day 42, Day 84
  At each time pion mentioned above, subjects will complete a Vaginal Symptoms questionnaire, subject will complete the questionnaire on their own.
Change in VMI (Vaginal Maturation Index) | Day 0, Day 14, Day 42
  At each time pion mentioned above, Cells will be collected to determine the vaginal maturation index.
Change in vaginal pH | Day 0, Day 14, Day 42
  At each time pion mentioned above, Vaginal pH will be determined
Change in pro-inflammatory cytokine levels in vaginal secretions | Day 0, Day 14, Day 42
  At each time pion mentioned above, vaginal secretions will be sampled by swab and samples will be frozen for determination of cytokine levels at a later time piont.

CONTACTS AND LOCATIONS:
Overall Officials: Gabe Nussbaum, MD, PhD, Study Director — Izun Pharma Ltd
Locations (3):
- United States (2):
  - Eastchester Medical Associates, The Bronx, New York
  - Seattle Women's, Seattle, Washington
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided